CLINICAL TRIAL: NCT05016401
Title: Multicenter Observational Study Evaluating the Performance and Safety of Use of the "KONTACT PERIO LEVEL" Dental Implant in Routine Clinical Practice.
Brief Title: Performance and Safety of Use of the "KONTACT PERIO LEVEL" Transgingival Titanium Dental Implant
Acronym: KPL
Status: Completed | Type: Observational
Sponsor: Biotech Dental (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-A01491-38
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2021-08

CONDITIONS: Tooth Loss; Partially Edentulous Maxilla; Partially Edentulous Mandible
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: KONTACT PERIO LEVEL (KPL) — The Kontact™ Perio Level is an implant with a transgingival neck that facilitates one-step surgery.

SUMMARY:
As part of post-marketing clinical follow-up, BIOTECH DENTAL sets up the collection and evaluation of clinical data proactively with the aim of confirming the safety, performance as well as the constantly acceptable nature of the risks identified and of detecting potential emerging risks with the use of "Kontact Perio Level" implants in everyday practice.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous patient requiring the placement of one (or more) dental implant (s) in the maxilla or mandibular
* Age ≥ 18 years old
* Good general health (ASA score between [1-2])
* Sufficient volume and bone quality (with or without bone graft) to support the implant
* Non-objection of the patient for the collection of his medical data as part of the study

Exclusion Criteria:

* Poor oral hygiene
* Bruxism, parafunctional habits, occlusion disorders and / or temporomandibular joints
* Infections and oral inflammation such as active periodontitis, active gingivitis
* Patient with metabolic disorders (eg diabetes mellitus) or bone disease that may compromise peri-implant tissue healing
* Heavy smoker (> 10 cigarettes / day)
* Patient with a pathology or immunosuppressive therapy such as chemotherapy, radiotherapy
* Patient on prolonged steroid therapy
* Titanium / titanium alloy allergy
* Alcohol or drug abuse
* Pregnant woman (or likely to be pregnant); or breastfeeding
* Difficulty of medical follow-up patients with geographical, social or psychological constraints
* Persons deprived of liberty or guardianship
* Involuntary / patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient eligible and planned for an implant-supported prosthetic restoration according to the instructions for use of the KONTACT PERIO LEVEL dental implant.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Success rate | 12 months
  For an implant to be declared "successful" it must meet the following criteria as defined by Albrektsson et al. 1986 adapted: Lack of mobility ; Absence of pain ; Lack of radiolucency around the implant ; Absence of bleeding and inflammation ; No significant peri-implant periodontal pocket (≤4mm) ; Stability of the peri-implant bone level over time with marginal bone loss ≤1.5 mm the first year and ≤0.2 mm the following years

SECONDARY OUTCOMES:
Bone Level | 12 months
  Peri-implant marginal bone loss and / or regrowth is calculated using x-rays
Prosthetic complications | 12 months
  All prosthetic complications having affected the restorations on implants, from the placement of the provisional restorations until the end of the study, are recorded (loosening of the abutment screws, the fracture of the abutment, loss of retention, fracture, etc.)
Primary stability | surgical time
  Value of the torque during implant placement
Survival rate | 12 months
  An implant is classified as "surviving" if it is still in operation at some point t
Factors that influence the survival and success rate | 12 months
  Univariate statistical analysis of the success and survival rate as a function of: age; sex; bone density; site of implantation; bone graft; type of prosthesis; jaw type;...
Peri-implantitis | 12 months
  Number of peri-implantitis (inflammatory disease causing bone loss around an implant)
Quality of Life | 12 months
  Evolution of the quality of life score calculated using GOHAI (General Oral Health Assessment Index)

CONTACTS AND LOCATIONS:
Locations (1):
- Coordinating Investigator, Bandol, France

IPD SHARING:
Plan to Share IPD: No